CLINICAL TRIAL: NCT01808521
Title: A Pilot Study of N-acetylcysteine in Suspected Thrombotic Thrombocytopenia Purpura
Brief Title: A Pilot Study of N-acetylcysteine in Thrombotic Thrombocytopenia Purpura
Acronym: NACinTTP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Bloodworks (Other)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N-Acetylcysteine in TTP
Record Dates: First submitted 2013-02-22; First posted 2013-03-11 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Purpura, Thrombotic Thrombocytopenic; TTP
Keywords: Purpura, Thrombotic Thrombocytopenic; TTP
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- N-acetylcysteine (Experimental): IV administration of N-acetylcysteine (Acetadote) at 150mg/Kg loading bolus over 60 minutes followed by 150mg/Kg over 17 hours if loading dose was well tolerated.
  Interventions: Drug: N-Acetylcysteine

INTERVENTIONS:
Drug: N-Acetylcysteine — IV administration of N-Acetylcysteine at 150mg/kg over 60 min first, then if well tolerated, 150mb/kg over 17 hours
  Other Names: Acetadote

SUMMARY:
In this study, the investigators want to determine if N-acetylcysteine(NAC), given intravenously, will decrease complications in patients with Thrombotic Thrombocytopenia Purpura (TTP) who are receiving treatment with therapeutic plasma exchange (TPE). The investigators want to determine, through anti-oxidant activity, if NAC will have additional efficacy in TTP by improving cleavage of the patients' VWF by ADAMTS13, and preventing propagation of platelet/VWF strings. This will be manifest by a more rapid improvement in the patient's platelet count, decrease in number of days requiring TPE, and decrease in microvascular thrombotic complications. The investigators will additionally: 1) Assess safety of NAC by evaluating subjects for adverse events and significant adverse events 2) Determine effects on TTP by measuring clinical and research laboratory values 3) Determine drug effects by measuring clinical and research laboratory values.

DETAILED DESCRIPTION:
Thrombotic thrombocytopenic purpura (TTP) is a rare hemostatic disorder with life threatening consequences secondary to microvascular thrombosis. While the use of therapeutic plasma exchange (TPE) has greatly improved survival, end organ damage, resistance to therapy, and relapses occur in many patients. Ultra-large von Willebrand factor multimers (ULVWF) are pathogenic in TTP. The investigators have found that N-acetylcysteine (NAC) cleaves ULVWF in vitro and in vivo in the ADAMTS13 deficient mice that are at increased risk of TTP. NAC is well tolerated in humans at intravenous doses used for treatment of acetaminophen overdose. This dosage correlates with that producing an effect in the murine studies noted above, and thus is an attractive treatment for patients with TTP. By cleaving VWF and preventing propagation of platelet/VWF strings, the investigators hypothesize that NAC treatment will decrease complications in patients with TTP receiving treatment with TPE. This will be manifest by a more rapid improvement in platelet count, decrease in number of days requiring plasma exchange, and decrease in microvascular thrombotic complications. To prepare for a larger trial the investigators propose a pilot study in 3 patients with suspected TTP at the University of Washington (UW) Medical Center. The study will be approved by the UW IRB prior to study initiation. Patients who consent to the study will receive daily NAC infusions beginning after the first TPE, in doses used for acetaminophen overdose. Blood samples will be collected for laboratory assays to determine optimal timing for sample collection in the larger multicenter trial, and to pilot the data collection forms. The investigators will also evaluate safety and patient tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years of age
2. Diagnosis of suspected TTP (lab evidence of hemolysis, platelet count <120,000, schistocytes on peripheral smear)
3. Plans for or just initiated therapeutic plasma exchange (TPE), and before 3rd TPE
4. Normal baseline prothrombin time (PT) and activated partial thromboplastin time (aPTT)
5. Anticipated TPE for > 5 days

Exclusion Criteria:

1. Asthma
2. Life expectancy < 1 week
3. Liver function tests abnormal- (ALT, direct bilirubin > three times upper normal limit)
4. Known underlying bleeding disorder
5. Pregnancy or nursing
6. Known allergy to NAC
7. Phosphodiesterase Type 5 inhibitors, nitroglycerin, or carbamazepine current use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-05; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Changes in platelet count | Daily for 7 days and at hospital discharge, expected to be at 1-2 weeks post infusion.
  The platelet count will be measured before, daily during 4 days of NAC infusion, the subsequent 3 days and on the day of hospital discharge which is estimated to be at 1-2 weeks post infusion. Changes in platelet count over time will be reported.

SECONDARY OUTCOMES:
Laboratory measures of VWF activity | Daily for 7 days and at hospital dischargewhich is estimated to be at 1-2 weeks post-infusion
  VWF levels, oxidation and activity will be measured before, each day of NAC infusion, the subsequent 3 days and at hospital discharge, expected to be at 1-2 weeks post-infusion. Changes in values over time will be reported.
Laboratory measures of ADAMTS13 activity | Daily for 7 days and at hospital discharge which is estimated to be at 1-2 weeks post-infusion
  ADAMTS13 level, oxidation and activity will be measured before, daily during the NAC infusion, for the 3 subsequent days and at hospital discharge, expected to be at 1-2 weeks post-infusion. Changes over time will be reported.
Laboratory measures of red blood cell (RBC) hemolysis and oxidation | Daily for 7 days and at hospital discharge which is estimated to be at 1-2 weeks post-infusion
  Laboratory markers of RBC hemolysis and oxidation will be measured before, daily during the NAC infusion, for 3 subsequent days and at hospital discharge, expected to be at 1-2 weeks post-infusion. Changes in values over time will be reported.
Safety of NAC infusion | Over the study period
  Adverse events will be collected daily during the hospitalization, at 2 weeks and 8 weeks following infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A Konkle, MD, Principal Investigator — Bloodworks
Locations (1):
- Puget Sound Blood Center, Seattle, Washington, United States